CLINICAL TRIAL: NCT00000978
Title: An Open-Label, Randomized, Dose-Finding, Multicenter Trial of Dideoxycytidine (ddC) Administered Concurrently With Zidovudine (AZT) in the Treatment of AIDS or Advanced ARC
Brief Title: A Study of Dideoxycytidine Plus Zidovudine in the Treatment of AIDS or Advanced AIDS Related Complex (ARC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Purpose: Treatment
Other Study IDs: ACTG 106; Protocol N3447
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 1992-08

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To determine the safety, tolerability, and activity of zidovudine (AZT) and zalcitabine (dideoxycytidine; ddC) and the bloodstream levels of these drugs in patients with AIDS or advanced AIDS-related complex (ARC).

Treatments using AZT alternating with ddC are being evaluated in ongoing trials with a goal of reducing the toxicity of each while maintaining antiviral effects. In addition, AZT and ddC may work together in a way that both drugs can be taken at lower doses or less frequent intervals when given together. If the doses can be reduced, then toxicity associated with long-term use of one drug may be reduced. Combination of AZT and ddC might reduce the likelihood of the emergence of resistant mutants. Recent studies indicate a reduced sensitivity of HIV isolated from patients after prolonged AZT therapy. Although the clinical significance of this finding is not clear, it would indicate that these combination studies are all the more important. HIV strains with decreased sensitivity to AZT are still sensitive to ddC.

DETAILED DESCRIPTION:
Treatments using AZT alternating with ddC are being evaluated in ongoing trials with a goal of reducing the toxicity of each while maintaining antiviral effects. In addition, AZT and ddC may work together in a way that both drugs can be taken at lower doses or less frequent intervals when given together. If the doses can be reduced, then toxicity associated with long-term use of one drug may be reduced. Combination of AZT and ddC might reduce the likelihood of the emergence of resistant mutants. Recent studies indicate a reduced sensitivity of HIV isolated from patients after prolonged AZT therapy. Although the clinical significance of this finding is not clear, it would indicate that these combination studies are all the more important. HIV strains with decreased sensitivity to AZT are still sensitive to ddC.

Patients are randomly assigned to one of six treatment groups of various dose combinations of AZT and ddC. Patients are evaluated every week for the first 10 weeks and biweekly thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine 300 mg per 4 weeks.
* Drugs unlikely to cause increased toxicity with either study drug and unlikely to cause peripheral neuropathy.
* Drugs with little nephrotoxicity, hepatotoxicity, or cytotoxicity, that patient has been taking and tolerating well for ongoing condition.
* Acyclovir (= or < 600 mg/day, orally).
* Ketoconazole (= or < 400 mg/day).
* Nystatin (occasional).
* Acetaminophen or nonsteroidal antiinflammatory agents (low dose).
* Drugs that could possibly cause serious additive toxicity when coadministered with either study drug, but unlikely to cause peripheral are allowed only if their use is anticipated for treatment of acute intercurrent illness or opportunistic infections.
* Allowed only with a study drug interruption of up to 21 days per episode, for a total of 42 days for the study:
* Acyclovir (> 600 mg/day).
* Experimental drugs including ganciclovir.
* Fluconazole.
* Systemic pentamidine.
* Pyrimethamine.
* Triple sulfa.
* Ansamycin.
* Prolonged continuous use of high-dose nonsteroidal antiinflammatory agents.
* Acetaminophen.
* Amphotericin.
* Foscarnet.

Concurrent Treatment:

Allowed:

* Radiation therapy if unlikely to cause peripheral neuropathy if their use is anticipated for treatment of acute intercurrent illness or opportunistic infection.
* Transfusion for anemia.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Active opportunistic infections requiring treatment with unallowed drugs.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within month prior to study entry, or with concurrent neoplasms other than KS, basal cell carcinoma of the skin, or in situ carcinoma of the cervix.
* History of peripheral neuropathy or any significant signs or symptoms of neurological disease, or abnormality indicative of peripheral neuropathy.
* Significant cardiac disease defined as history of ventricular arrhythmias requiring medication, prior myocardial infarction, or history of angina or ischemic changes on electrocardiogram.
* Significant liver disease as defined by transaminase levels or by history of cirrhosis or ascites.
* Significant renal disease defined by serum creatinine.

Concurrent Medication:

Excluded:

* Experimental drugs including fluconazole, and foscarnet.
* Immunomodulators including interferon, interleukins, or systemic corticosteroids.
* Ganciclovir.
* Neurotoxic drugs.
* Drugs that could potentially cause peripheral neuropathy, including chloramphenicol, cisplatin, iodoquinol, dapsone, phenytoin, disulfiram, ethionamide, glutethimide, gold, hydralazine, isoniazid, metronidazole, vincristine, and nitrofurantoin.
* Excluded within 4 weeks of study entry:
* Drugs that have caused significant nephrotoxicity or significant hepatotoxicity (as defined by transaminases).

Concurrent Treatment:

Excluded:

* Transfusion dependent.

Patients are excluded if unwilling or unable to sign informed consent.

Prior Medication:

Excluded:

* Zidovudine (AZT).
* Dideoxycytidine (ddC).
* Any other nucleoside antiretrovirals.

Positive antibody to HIV using any federally licensed ELISA test kit. Diagnosis of AIDS or AIDS-related complex (ARC).

Active substance or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of Miami School of Medicine, Miami, Florida

REFERENCES:
- [Background] Meng TC, Fischl MA, Boota AM, Spector SA, Bennett D, Bassiakos Y, Lai SH, Wright B, Richman DD. Combination therapy with zidovudine and dideoxycytidine in patients with advanced human immunodeficiency virus infection. A phase I/II study. Ann Intern Med. 1992 Jan 1;116(1):13-20. doi: 10.7326/0003-4819-116-1-13. PMID 1345755
- [Background] Meng TC, Boota A, Fischl MA, Spector SA, McCaan M, Richman DD. ACTG 106: Phase I/II dose finding study of concurrently administered dideoxycytidine (ddC) and zidovudine (ZDV, AZT). Int Conf AIDS. 1990 Jun 20-23;6(3):192 (abstract no SB426)
- [Background] Meng TC, Fischl MA, Richman DD. AIDS Clinical Trials Group: phase I/II study of combination 2',3'-dideoxycytidine and zidovudine in patients with acquired immunodeficiency syndrome (AIDS) and advanced AIDS-related complex. Am J Med. 1990 May 21;88(5B):27S-30S. doi: 10.1016/0002-9343(90)90419-e. PMID 2159707
- [Background] Gries JM, Troconiz IF, Verotta D, Jacobson M, Sheiner LB. A pooled analysis of CD4 response to zidovudine and zalcitabine treatment in patients with AIDS and AIDS-related complex. Clin Pharmacol Ther. 1997 Jan;61(1):70-82. doi: 10.1016/S0009-9236(97)90183-1. PMID 9024175